CLINICAL TRIAL: NCT02438826
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Study of : Galcanezumab (LY2951742) With a Long-Term Open-Label Extension in Patients With Chronic Cluster Headache
Brief Title: A Study of Galcanezumab in Participants With Chronic Cluster Headache
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15781; I5Q-MC-CGAM (Other: Eli Lilly and Company); 2014-005429-11 (EudraCT Number)
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-06

CONDITIONS: Chronic Cluster Headache
MeSH Terms: conditions — Cluster Headache | interventions — galcanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Galcanezumab 300 mg (Experimental): Double-Blind Treatment Phase: Participants received galcanezumab 300 mg once a month by subcutaneous (SC) injection for 3 months.
  Open-Label Treatment Phase: Participants received 300 mg galcanezumab by subcutaneous injections every 30 days, for up to a total of 12 administrations.
  Interventions: Drug: Galcanezumab 300 mg
- Placebo (Placebo Comparator): Double-Blind Treatment Phase: Participants received placebo once a month by subcutaneous (SC) injection for 3 months.
  Open-Label Treatment Phase: Participants received 300 mg galcanezumab by subcutaneous injections every 30 days, for up to a total of 12 administrations.
  Interventions: Drug: Galcanezumab 300 mg; Drug: Placebo

INTERVENTIONS:
Drug: Galcanezumab 300 mg — Administered SC
  Other Names: LY2951742
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy of the study drug known as galcanezumab in participants with chronic cluster headache.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a history of chronic cluster headache occurring without a remission period, or with remissions lasting <1 month, for at least 1 year.
* Participants are able to distinguish cluster headache attacks from other headaches.

Exclusion Criteria:

* Current enrollment in or discontinuation within the last 30 days from, a clinical trial involving any investigational drug or device.
* Current use or any prior exposure to any calcitonin-gene-related peptide (CGRP) antibody, any antibody to the CGRP receptor, or antibody to nerve growth factor (NGF).
* Are taking indomethacin and/or are suspected of having another distinct trigeminal autonomic cephalalgia.
* A history of migraine variants that could implicate or could be confused with ischemia.
* Known hypersensitivity to multiple drugs, monoclonal antibodies or other therapeutic proteins.
* A history or presence of other medical illness that indicates a medical problem that would preclude study participation.
* Evidence of significant active or unstable psychiatric disease, in the opinion of the investigator.
* Women who are pregnant or nursing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2015-06-18 (Actual); Primary Completion 2018-03-27 (Actual); Study Completion 2019-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (46):
- United States (13):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - California Medical Clinic for Headache, Santa Monica, California
  - Stanford University Hospital, Stanford, California
  - Colorado Neurological Institute, Englewood, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - New England Institute for Clinical Research, Stamford, Connecticut
  - Mayo Clinic-Jacksonville, Jacksonville, Florida
  - Tampa General Hospital, Tampa, Florida
  - Michigan Head, Pain and Neurological Institute, Ann Arbor, Michigan
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Southwestern Medical Center - Dallas, Dallas, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
- Belgium (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Ghent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Liège
- Canada (3):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Montreal
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Toronto
- Denmark (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glostrup Municipality
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Glostrup Municipality
- Finland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Helsinki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Turku
- France (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Nice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Etienne
- Germany (6):
  - Praxis Dr. Stude, Bochum
  - Universtitätsklinikum Essen AöR, Essen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Jena
  - Migräne- und Kopfschmerzklinik GmbH & Co. KG, Königstein
  - Klinikum der Universität München Campus Großhadern, München
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Athens, Greece
- Italy (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Florence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Pavia
- Netherlands (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Nijmegen
- Spain (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Valencia
- United Kingdom (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Hull
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Liverpool
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Jensen RH, Tassorelli C, Myers Oakes TM, Bardos JN, Zhou C, Dong Y, Aurora SK, Martinez JM. Baseline demographics and disease characteristics of patients with episodic or chronic cluster headache: data from two phase 3 randomized clinical trials in Europe and North America. Front Neurol. 2023 Dec 15;14:1293163. doi: 10.3389/fneur.2023.1293163. eCollection 2023. PMID 38162453
- [Derived] Dodick DW, Goadsby PJ, Lucas C, Jensen R, Bardos JN, Martinez JM, Zhou C, Aurora SK, Yang JY, Conley RR, Oakes T. Phase 3 randomized, placebo-controlled study of galcanezumab in patients with chronic cluster headache: Results from 3-month double-blind treatment. Cephalalgia. 2020 Aug;40(9):935-948. doi: 10.1177/0333102420905321. Epub 2020 Feb 12. PMID 32050782
- See also: Click here for more information about this study: A Study of LY2951742 in Participants With Chronic Cluster Headache — http://www.lillytrialguide.com/EN-us/studies/headache/cgam

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study consists of a 12-week double-blind treatment phase; an optional 1-year open-label treatment phase; and a 16-week post-treatment phase (washout).
Groups:
- Placebo/Galcanezumab (GMB) 300 mg: Double-Blind Treatment Phase: Participants received placebo once a month by subcutaneous (SC) injection for 3 months.
  Open-Label Treatment Phase: Participants from placebo group received 300 milligrams (mg) of galcanezumab (GMB) by subcutaneous injection every 30 days, for up to a total of 12 administrations.
  Post-Treatment Phase: Participants from Open-Label Treatment Phase entered this phase, they have not received any intervention during this post-treatment period.
- GMB 300 mg/GMB 300 mg: Double-Blind Treatment Phase: Participants received galcanezumab 300 mg once a month by subcutaneous (SC) injection for 3 months.
  Open-Label Treatment Phase: Participants from galcanezumab group received 300 mg of galcanezumab by subcutaneous injection every 30 days, for up to a total of 12 administrations.
  Post-Treatment Phase: Post-Treatment Phase: Participants from Open-Label Treatment Phase entered this phase, they have not received any intervention during this post-treatment period.
- Placebo (Post-Treatment Phase); Galcanezumab 300 mg (Post-Treatment Phase): Participants from double blind treatment group entered this phase, they have not received any intervention during this post-treatment period.
Period: Double-Blind Treatment Phase
Arm/Group | Placebo/Galcanezumab (GMB) 300 mg | GMB 300 mg/GMB 300 mg | Placebo (Post-Treatment Phase) | Galcanezumab 300 mg (Post-Treatment Phase)
Started | 123 | 117 | 0 | 0
Received at Least 1 Dose of Study Drug | 120 | 117 | 0 | 0
Completed | 117 | 113 | 0 | 0
Not Completed | 6 | 4 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 0 | 0
Not completed — Screen Failure | 2 | 0 | 0 | 0
Period: Open-Label Treatment Phase
Arm/Group | Placebo/Galcanezumab (GMB) 300 mg | GMB 300 mg/GMB 300 mg | Placebo (Post-Treatment Phase) | Galcanezumab 300 mg (Post-Treatment Phase)
Started | 116 (This period is optional phase, one participant chose not to enter the open-label phase.) | 113 | 0 | 0
Completed | 72 | 80 | 0 | 0
Not Completed | 44 | 33 | 0 | 0
Not completed — Adverse Event | 11 | 6 | 0 | 0
Not completed — Lack of Efficacy | 27 | 18 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 7 | 0 | 0
Period: Post-Treatment Phase
Arm/Group | Placebo/Galcanezumab (GMB) 300 mg | GMB 300 mg/GMB 300 mg | Placebo (Post-Treatment Phase) | Galcanezumab 300 mg (Post-Treatment Phase)
Started | 93 (Participants who discontinued Open-Label Treatment also had the option to enter Post-Treatment Phase) | 93 (Participants who discontinued Open-Label Treatment also had the option to enter Post-Treatment Phase) | 2 (Participants entered from Double-Blind Treatment Phase.) | 4 (Participants entered from Double-Blind Treatment Phase.)
Completed | 84 | 92 | 2 | 4
Not Completed | 9 | 1 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 0
Not completed — Lack of Efficacy | 4 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Placebo: Participants received placebo once a month by subcutaneous (SC) injection for 3 months.
- Galcanezumab 300 mg: Participants received galcanezumab 300 mg once a month by subcutaneous (SC) injection for 3 months.
- Total: Total of all reporting groups
Arm/Group | Placebo | Galcanezumab 300 mg | Total
Number analyzed (Participants) | 120 | 117 | 237
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.38 (10.81) | 45.62 (11.03) | 45.00 (10.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 31 | 65
  Male | 86 | 86 | 172
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 18 | 33
  Not Hispanic or Latino | 87 | 81 | 168
  Unknown or Not Reported | 18 | 18 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 101 | 99 | 200
  More than one race | 18 | 17 | 35
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Greece | 0 | 1 | 1
  Canada | 4 | 4 | 8
  Netherlands | 5 | 5 | 10
  Belgium | 16 | 16 | 32
  United States | 15 | 18 | 33
  Finland | 2 | 2 | 4
  Denmark | 5 | 4 | 9
  Italy | 17 | 14 | 31
  United Kingdom | 8 | 8 | 16
  France | 20 | 20 | 40
  Germany | 22 | 20 | 42
  Spain | 6 | 5 | 11
Weekly Cluster Headache Attacks [Mean (Standard Deviation); unit: cluster headache attacks per week] | 18.47 (10.66) | 19.18 (9.82) | 18.82 (10.24)
Lifetime Suicidal Ideation Prior to Screening [Count of Participants; unit: Participants] — Suicidal ideation was defined as a "yes" answer to any 1 of 5 suicidal ideation questions, which included = Wish to be Dead; Non-specific Active Suicidal Thoughts; Active Suicidal Ideation with Any Methods (No Plan); Active Suicidal Ideation with Some Intent to Act, without a Specific Plan; Active Suicidal Ideation with Intent to Act.
  Participants | 30 | 25 | 55
Lifetime Suicidal Behavior Prior to Screening [Count of Participants; unit: Participants] — Suicidal behavior was defined as a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt (non-fatal), and completed suicide. Population: All randomized participants who received at least 1 dose of study drug and had a baseline value for Lifetime Suicidal Behavior.
  Participants
    number analyzed (Participants) | 119 | 117 | 236
    (all) | 5 | 4 | 9
Verapamil Use at Baseline [Count of Participants; unit: Participants] | 63 | 55 | 118

OUTCOME MEASURES:

1. Primary Outcome: Overall Mean Change From Baseline in Weekly Cluster Headache Attack Frequency
Description: Number of cluster headache attacks was recorded daily by study participants in their ePRO Diary, Baseline and 12 weeks of daily data during double-blind treatment phase will be converted into 14-calendar day intervals: the baseline 14-day interval, Weeks 1/2, 3/4, 5/6, 7/8, 9/10, and 11/12. Next, the biweekly interval results were adjusted to 7-day (weekly) interval in order to report the outcome as weekly frequency. Overall mean change from baseline is derived from mixed model repeated measures (MMRM) analysis. Least Square (LS) means were calculated using MMRM model with treatment, sex, verapamil use, pooled investigative site, week, baseline, and treatment by week as fixed effects.
Time Frame: Baseline, Week 1 through Week 12
Population: All randomized participants who received at least 1 dose of study drug, and had baseline and at least one post baseline value.
Measure: Least Squares Mean (Standard Error); unit: cluster headache attacks per week
Arm/Group | Placebo | Galcanezumab 300 mg
Number analyzed (Participants) | 120 | 117
cluster headache attacks per week | -4.59 (0.79) | -5.38 (0.81)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 300 mg; Test type: Superiority; p = 0.334, Mixed Models Analysis — Cui, Hung, Wang (CHW) procedure applied; LSMean Difference = -0.80, 95% CI 2-sided [-2.77 to 1.17]

2. Secondary Outcome: Percentage of Participants With a 50% or Greater Reduction From Baseline in the Weekly Number of Cluster Headache Attacks
Description: A 50% responder is any participant who has a ≥50% reduction from baseline in the weekly number of cluster headache attacks in a 14-day interval: Weeks 1/2, Weeks 3/4, Weeks 5/6, Weeks 7/8, Weeks 9/10, and Weeks 11/12. Mean percentage of participants is derived from the average of weeks 1/2 to weeks 11/12 from generalized linear mixed model repeated measures method with treatment, sex, verapamil use, week, treatment by week, and baseline as fixed effects.
Time Frame: Baseline, Week 1 through Week 12
Population: All randomized participants who received at least 1 dose of study drug, and had baseline and at least 1 post baseline value.
Measure: Mean (Standard Error); unit: percentage of participants
Arm/Group | Placebo | Galcanezumab 300 mg
Number analyzed (Participants) | 120 | 117
percentage of participants | 27.1 (3.5) | 32.6 (3.8)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 300 mg; Test type: Superiority; p = 0.170, Mixed Models Analysis — Cui, Hung, Wang (CHW) procedure applied; Odds Ratio (OR) = 1.297, 95% CI 2-sided [0.830 to 2.028]

3. Secondary Outcome: Percentage of Participants With a Sustained Response of 50% or Greater Reduction From Baseline in the Weekly Number of Cluster Headache Attacks
Description: Sustained Response is defined as a 50% or greater reduction in the weekly cluster attack frequency from baseline to Weeks 3/4 and maintained at Weeks 5/6, Weeks 7/8, Weeks 9/10, and Weeks 11/12. Percentage of participants with a sustained response was analyzed using Koch's nonparametric randomization-based analysis of covariance method. This method adjusted for pooled investigative site by including it as a stratification variable. It also adjusted for sex, verapamil use and baseline value.
Time Frame: Baseline, Week 3 through Week 12
Population: All randomized participants who received at least 1 dose of study drug, had a baseline, and at least one post baseline value.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Galcanezumab 300 mg
Number analyzed (Participants) | 120 | 117
percentage of participants | 17.50 | 16.24
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 300 mg; Test type: Superiority; p = 0.946, Mixed Models Analysis — Chui, Hung, Wang (CHW) procedure applied)

4. Secondary Outcome: Percentage of Participants With a 30% Reduction in the Weekly Number of Cluster Headache Attacks
Description: A 30% responder is any participant who has a ≥30% reduction from baseline in the weekly number of cluster headache attacks in a 14-day interval. Weeks 1/2, 3/4, 5/6, 7/8, 9/10, and 11/12. Mean percentage of participants is derived from the average of weeks 1/2 to weeks 11/12 from generalized linear mixed model repeated measures method with treatment, sex, verapamil use, week, treatment by week, and baseline as fixed effects. .
Time Frame: Baseline, Week 1 through Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percentage of participants
Arm/Group | Placebo | Galcanezumab 300 mg
Number analyzed (Participants) | 120 | 117
percentage of participants | 39.0 (3.9) | 49.1 (4.1)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 300 mg; Test type: Superiority; p = 0.057, Mixed Models Analysis; Odds Ratio (OR) = 1.510, 95% CI 2-sided [0.987 to 2.309]

5. Secondary Outcome: Percentage of Participants Reporting a Score of 1 or 2 on the Patient Global Impression of Improvement (PGI-I)
Description: PGI-I requests participants to mark the box that best describes their cluster headache condition since they started taking the medicine. The options in the displayed boxes are represented on a 7-point scale, with 1 = very much better, 2 = much better, 3 = a little better, 4 = no change, 5 = a little worse, 6 = much worse, and 7 = very much worse. Percentage of participants were derived with a generalized linear mixed model repeated measures method with treatment, sex, verapamil use, baseline cluster headache attack category, month, and treatment by month as fixed effects.
Time Frame: Week 4
Population: All randomized participants who received at least one dose of study drug and had PGI-I measurement at Week 4.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Galcanezumab 300 mg
Number analyzed (Participants) | 92 | 88
percentage of participants | 19.4 | 21.5
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 300 mg; Test type: Superiority; p = 0.713, Mixed Models Analysis; Odds Ratio (OR) = 1.141, 95% CI 2-sided [0.563 to 2.314]

6. Secondary Outcome: Percentage of Participants Reporting a Score of 1 or 2 on the Patient Global Impression of Improvement (PGI-I)
Description: as for outcome 5
Time Frame: Week 8
Population: All randomized participants who received at least one dose of study drug and had PGI-I measurement at Week 8.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Galcanezumab 300 mg
Number analyzed (Participants) | 97 | 86
percentage of participants | 32.0 | 32.1
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 300 mg; Test type: Superiority; p = 0.979, Mixed Models Analysis; Odds Ratio (OR) = 1.008, 95% CI 2-sided [0.548 to 1.856]

7. Secondary Outcome: Percentage of Participants Reporting a Score of 1 or 2 on the Patient Global Impression of Improvement (PGI-I)
Description: as for outcome 5
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study drug and had PGI-I measurement at week 12.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Galcanezumab 300 mg
Number analyzed (Participants) | 95 | 95
percentage of participants | 35.6 | 30.4
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 300 mg; Test type: Superiority; p = 0.437, Mixed Models Analysis; Odds Ratio (OR) = 0.788, 95% CI 2-sided [0.431 to 1.440]

8. Secondary Outcome: Percentage of Participants With Suicidal Ideation Assessed by Columbia - Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. The scale includes suggested questions to solicit the type of information needed to determine if a suicide-related thought or behavior occurred. Some questions are binary responses (yes/no) and some are on a scale of 1 (low severity) to 5 (high severity). Suicidal ideation: a "yes" answer to any of 5 suicidal ideation questions: wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods without intent to act, active suicidal ideation with some intent to act without specific plan, active suicidal ideation with specific plan and intent.
Time Frame: Week 1 through Week 12
Population: All randomized participants who received at least one dose of study drug and had at least one post baseline C-SSRS assessment.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Placebo administered by SQ injection every 30 Days for 12 weeks.
- Galcanezumab 300 mg: 300 mg galcanezumab (LY2951742) administered by subcutaneous (SQ) injection every 30 days for 12 weeks.
Arm/Group | Placebo | Galcanezumab 300 mg
Number analyzed (Participants) | 119 | 116
percentage of participants | 5.04 | 4.31

9. Secondary Outcome: Percentage of Participants With Suicidal Behaviors Assessed by Columbia - Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. The scale includes suggested questions to solicit the type of information needed to determine if a suicide-related thought or behavior occurred. Some questions are binary responses (yes/no) and some are on a scale of 1 (low severity) to 5 (high severity). Suicidal behavior: a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide.
Time Frame: Week 1 through Week 12
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Galcanezumab 300 mg
Number analyzed (Participants) | 119 | 116
percentage of participants | 0 | 0

10. Secondary Outcome: Percentage of Participants Developing Anti-Drug Antibodies (ADA) to Galcanezumab (LY2951742)
Description: Treatment emergent (TE) ADA evaluable participant is considered to be TE ADA+ if the subject has at least one post-baseline titer that is a 4-fold or greater increase in titer from baseline measurement. If baseline result is ADA Not Present, then the participant is TE ADA+ if there is at least one post-baseline result of ADA present with titer >= 1: 20.
Time Frame: Baseline, Week 1 through Week 12
Population: All randomized participants who received at least one dose of study drug and had non-missing baseline ADA result, and at least one non-missing post baseline ADA result.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Galcanezumab 300 mg
Number analyzed (Participants) | 115 | 113
percentage of participants | 0 | 0.88

11. Secondary Outcome: Pharmacokinetics (PK): Serum Concentration of Galcanezumab
Description: Pharmacokinetics (PK): Serum Concentration of Galcanezumab
Time Frame: Week 2
Population: All randomized participants who received at least 1 dose of study drug and had evaluable galcanezumab PK samples at Week 2.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Galcanezumab 300 mg
Number analyzed (Participants) | 90
nanogram per milliliter | 30,600 (10,700)

12. Secondary Outcome: Pharmacokinetics (PK): Serum Concentration of Galcanezumab
Description: Pharmacokinetics (PK): Serum Concentration of Galcanezumab
Time Frame: Week 4
Population: All randomized participants who received at least 1 dose of study drug and had evaluable galcanezumab PK samples at Week 4.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Galcanezumab 300 mg
Number analyzed (Participants) | 96
nanogram per milliliter | 20,200 (6780)

13. Secondary Outcome: Pharmacokinetics (PK): Serum Concentration of Galcanezumab
Description: Pharmacokinetics (PK): Serum Concentration of Galcanezumab
Time Frame: Week 8
Population: All randomized participants who received at least 1 dose of study drug and had evaluable galcanezumab PK samples at Week 8.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Galcanezumab 300 mg
Number analyzed (Participants) | 94
nanogram per milliliter | 29,700 (11,500)

14. Secondary Outcome: Pharmacokinetics (PK): Serum Concentration of Galcanezumab
Description: Pharmacokinetics (PK): Serum Concentration of Galcanezumab
Time Frame: Week 12
Population: All randomized participants who received at least 1 dose of study drug and had evaluable galcanezumab PK samples at Week 12.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Galcanezumab 300 mg
Number analyzed (Participants) | 96
nanogram per milliliter | 31,100 (11,900)

ADVERSE EVENTS:
Time Frame: Up to 1 Year 7 Months
Description: All randomized participants who received at least 1 dose of study drug. Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Placebo (Double-Blind Treatment Phase): Participants received placebo once a month by subcutaneous (SC) injection for 3 months.
- Galcanezumab 300 mg (Double-Blind Treatment Phase): Participants received galcanezumab 300 mg once a month by subcutaneous (SC) injection for 3 months
- Placebo/GMB 300 mg (Open-Label Treatment Phase): Participants from placebo group received 300 mg of galcanezumab by subcutaneous injection every 30 days, for up to a total of 12 administrations.
- GMB 300 mg/GMB 300 mg (Open-Label Treatment Phase): Participants from galcanezumab of double-blind group received 300 mg of galcanezumab by subcutaneous injection every 30 days, for up to a total of 12 administrations.
- Placebo/GMB 300 mg (Post-Treatment Phase); GMB 300 mg/GMB 300 Mg-Post-Treatment Phase: Participants from Open-Label Treatment Phase entered this phase, they have not received any intervention during this post-treatment period.
Arm/Group | Placebo (Double-Blind Treatment Phase) | Galcanezumab 300 mg (Double-Blind Treatment Phase) | Placebo/GMB 300 mg (Open-Label Treatment Phase) | GMB 300 mg/GMB 300 mg (Open-Label Treatment Phase) | Placebo (Post-Treatment Phase) | Galcanezumab 300 mg (Post-Treatment Phase) | Placebo/GMB 300 mg (Post-Treatment Phase) | GMB 300 mg/GMB 300 Mg-Post-Treatment Phase
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/117 | 0/116 | 0/113 | 0/2 | 0/4 | 0/93 | 0/93
Serious Adverse Events (participants affected / at risk) | 3/120 | 2/117 | 11/116 | 10/113 | 0/2 | 0/4 | 0/93 | 5/93
Other Adverse Events (participants affected / at risk) | 60/120 | 68/117 | 69/116 | 72/113 | 1/2 | 2/4 | 18/93 | 16/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Double-Blind Treatment Phase) (N=120) | Galcanezumab 300 mg (Double-Blind Treatment Phase) (N=117) | Placebo/GMB 300 mg (Open-Label Treatment Phase) (N=116) | GMB 300 mg/GMB 300 mg (Open-Label Treatment Phase) (N=113) | Placebo (Post-Treatment Phase) (N=2) | Galcanezumab 300 mg (Post-Treatment Phase) (N=4) | Placebo/GMB 300 mg (Post-Treatment Phase) (N=93) | GMB 300 mg/GMB 300 Mg-Post-Treatment Phase (N=93)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amaurosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site urticaria (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cluster headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reversible cerebral vasoconstriction syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pregnancy of partner (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthrodesis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (Double-Blind Treatment Phase) (N=120) | Galcanezumab 300 mg (Double-Blind Treatment Phase) (N=117) | Placebo/GMB 300 mg (Open-Label Treatment Phase) (N=116) | GMB 300 mg/GMB 300 mg (Open-Label Treatment Phase) (N=113) | Placebo (Post-Treatment Phase) (N=2) | Galcanezumab 300 mg (Post-Treatment Phase) (N=4) | Placebo/GMB 300 mg (Post-Treatment Phase) (N=93) | GMB 300 mg/GMB 300 Mg-Post-Treatment Phase (N=93)
Palpitations (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 6 (8) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 1 (1) | 5 (6) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (8) | 6 (7) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 7 (9) | 5 (5) | 6 (6) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 5 (8) | 4 (4) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 1 (1) | 8 (11) | 5 (6) | 2 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 11 (15) | 14 (32) | 16 (32) | 8 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 7 (10) | 5 (7) | 2 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (2) | 8 (20) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (7) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (3) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2) | 4 (5) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 3 (4) | 2 (2) | 8 (8) | 5 (5) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Nasopharyngitis (Infections and infestations) | 15 (16) | 12 (13) | 14 (19) | 17 (24) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0/34 (0) | 0/31 (0) | 1/33 (1) | 0/29 (0) | 0/1 (0) | 0/2 (0) | 0/25 (0) | 0/25 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 5 (6) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) | 4 (4) | 10 (12) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 4 (4) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 6 (7) | 5 (5) | 4 (5) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 2 (3) | 2 (2) | 3 (6) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 5 (6) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 1 (1) | 2 (4) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/34 (0) | 1/31 (1) | 1/33 (1) | 0/29 (0) | 0/1 (0) | 0/2 (0) | 0/25 (0) | 0/25 (0)
Menstrual disorder (Reproductive system and breast disorders) | 0/34 (0) | 1/31 (1) | 0/33 (0) | 0/29 (0) | 0/1 (0) | 0/2 (0) | 0/25 (0) | 0/25 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0/34 (0) | 0/31 (0) | 0/33 (0) | 1/29 (1) | 0/1 (0) | 0/2 (0) | 0/25 (0) | 0/25 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0/34 (0) | 0/31 (0) | 0/33 (0) | 0/29 (0) | 0/1 (0) | 0/2 (0) | 1/25 (3) | 0/25 (0)
Hypertension (Vascular disorders) | 3 (3) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/26/NCT02438826/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT02438826/SAP_001.pdf